CLINICAL TRIAL: NCT00924742
Title: A Single-Dose Pharmacokinetics Study of Tapimycin Injection(Piperacillin 4 g + Tazobactam 0.5 g Powder for Injection) Administered Under Fasting Conditions to Healthy Adult Subjects
Brief Title: A Single-Dose Pharmacokinetics Study of Tapimycin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Feng-Yee Chang/The Head of Department of Internal Medicine, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MCPEM08026M1; 097-05-160; C163
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: The PK of Tapimycin; volunteer
MeSH Terms: interventions — Piperacillin; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test drug (Experimental)
  Interventions: Drug: Tapimycin (piperacillin 4 g + tazobactam 0.5g)

INTERVENTIONS:
Drug: Tapimycin (piperacillin 4 g + tazobactam 0.5g) — One intravenous infusion (piperacillin 4 g + tazobactam 0.5 g powder for injection) over 30 minutes/single dosing

SUMMARY:
The purpose of this study is to examine the pharmacokinetic properties of Tapimycin injection (piperacillin 4 g + tazobactam 0.5 g powder for injection) in healthy volunteers under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent before enrollment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
2. Healthy adult male, aged between 20 and 40 years old.
3. Body Mass Index (BMI) between 18.5 and 25.
4. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest x-ray and electrocardiogram.
5. No significant deviation from normal biochemistry.
6. No significant deviation from normal hematology.
7. No significant deviation from normal urinalysis.

Exclusion Criteria:

1. History of drug or alcohol abuse within the past year.
2. Medical history of severe drug allergy or sensitivity to analogous drug.
3. Acute or chronic diseases or having undergone surgery from 4 weeks prior to PeriodI dosing.
4. Any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology.
5. Ongoing peptic ulcer and constipation.
6. Planned vaccination during the time course of the study.
7. Taking any clinical study drug from 3 months prior to Period I dosing.
8. Use of any medication, including herb medicine or vitamins from 4 weeks before the study.
9. Blood donation of more than 500 mL within the past 3 months.
10. A positive Hepatitis B surface antigen or positive Hepatitis C antibody.
11. A positive test for HIV antibody.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To examine the pharmacokinetic properties | 8.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Yee Chang, Principal Investigator — Tri-Service General Hospital